CLINICAL TRIAL: NCT04357795
Title: Effect of Cequa™ in Subjects With Dry Eye Disease That Is Currently Inadequately Controlled While on Cyclosporine 0.05% Ophthalmic Emulsion
Brief Title: Effect of Cequa™ in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTX101-2019-001
Record Dates: First submitted 2020-04-08; First posted 2020-04-22 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-10

CONDITIONS: Dry Eye Disease
Keywords: Keratoconjunctivitis Sicca; KCS; Dry eye
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Cyclosporine; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CequaTM (Cyclosporine 0.09%) ophthalmic solution (Experimental)
  Interventions: Drug: CequaTM (Cyclosporine 0.09%) ophthalmic solution

INTERVENTIONS:
Drug: CequaTM (Cyclosporine 0.09%) ophthalmic solution — One drop CequaTM (Cyclosporine 0.09%) ophthalmic solution in each eye twice daily, approximately 12 hours apart.

SUMMARY:
This is a Phase 4, multicenter, single arm, 12 week study in subjects with dry eye disease, which is inadequately controlled by cyclosporine 0.05% ophthalmic emulsion.

DETAILED DESCRIPTION:
This is a phase 4, multicenter, open-label, single-arm, 12-week study of subjects with dry eye disease that is inadequately controlled by cyclosporine (CsA) 0.05% ophthalmic emulsion. Subject enrollment will be classified by evidence of dry eye disease (ie, signs, symptoms, or both signs and symptoms). Treatment will be one drop of CsA 0.09% ophthalmic solution (Cequa) in each eye twice daily (BID) for 12 weeks. The study hypothesis is that CsA 0.09% ophthalmic solution will show improved clinical benefit in subjects whose dry eye signs and/or symptoms are inadequately controlled while on CsA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with a history of bilateral dry eye disease for a period of at least 3 months.
2. Aged of at least 18 years.
3. Subjects with total corneal fluorescein staining ≥6 or corneal fluorescein staining in an individual zone ≥2 as per National Eye Institute Grading Scale.
4. Subjects with modified symptom assessment in dry eye global symptom score, ≥40 using visual analogue scale.
5. Subjects with best-corrected visual acuity 20/200 or better in both eyes at the Screening/Baseline visit

Exclusion Criteria:

1. Subjects who have used cyclosporin 0.05% ophthalmic emulsion in both eyes for less than 3 months prior to the Screening/Baseline visit.
2. Subjects with history of treatment failure with cyclosporin 0.05% ophthalmic emulsion.
3. Subjects who have active seasonal and/or perennial allergic conjunctivitis in either eye.
4. Subjects who had already Use initiated any systemic or topical ocular medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Eye Associates of Fort Myers, 4225 Evans Ave., Fort Myers, Florida
  - Bowden Eye and Associates, 7205 Bonneval Road, Jacksonville, Florida
  - Eye Center of N Florida, 2500 Martin Luther King Jr Blvd, Panama City, Florida
  - Kannarr Eye Care, 2521 N Broadway, Pittsburg, Kansas
  - Texas Eye and Laser Center, 1872 Norwood Dr. #200, Hurst, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Started | 134
Completed | 115
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 125
Age, Continuous [Mean (Full Range); unit: years] | 65.5 [23 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 107
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Baseline in Total Corneal Fluoroscein Staining Score
Description: Scale for Corneal Staining as defined by the FDA/NEI: 0-4 (0-no staining, 4-severe staining). The higher number indicates more severe. The lower the number indicates less severe staining on the cornea
Time Frame: Week12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 125
score on a scale | -3.1 (2.88)
Statistical Analysis 1: Comparison: CequaTM (Cyclosporine 0.09%) Ophthalmic Solution; Test type: Other — Single group analysis; p < 0.0001, Paired t-test

2. Primary Outcome: Change From Baseline in Modified Dry Eye Scoring.
Description: Based on questionnaire asked to subjects (sign and symptoms), modified symptom of dry eye score (range 0 to 100) will be assessed. Increase in score will indicate severity in the symptoms.
Time Frame: Week12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 125
score on a scale | -29.14 (26.220)
Statistical Analysis 1: Comparison: CequaTM (Cyclosporine 0.09%) Ophthalmic Solution; Test type: Other — Single group analysis; p < 0.0001, Paired t-test

3. Secondary Outcome: Mean Change in Baseline for Conjunctival Staining Assessment
Description: Based on Investigator's judgement, 6 areas of the conjunctiva will be evaluated in a low to moderate intensity.
  Scale for Conjunctival Staining defined: 0-6 (0 no staining, 6-severe staining). The higher the number indicates more severe. The lower the number indicates less severe staining on the conjunctival
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 124
score on a scale | -2.35 (2.918)
Statistical Analysis 1: Comparison: CequaTM (Cyclosporine 0.09%) Ophthalmic Solution; Test type: Other — Single group analysis; p < 0.0001, Paired t-test

4. Secondary Outcome: Changes From Baseline in Central Corneal Staining Score
Description: Five areas of cornea will be evaluated on a 0 to 4 scale and value from 0 (absent) to 4 (severe) to each section will be allotted based on NEI grading scale
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 125
score on a scale | -0.5 (0.87)
Statistical Analysis 1: Comparison: CequaTM (Cyclosporine 0.09%) Ophthalmic Solution; Test type: Other — Single group analysis; p < 0.0001, Paired t-test

5. Secondary Outcome: Mean Change in Baseline for Tear Osmolarity Score for Both Eyes
Description: Tear osmolarity of both the eyes will be assessed and score (mOsm/L) will be allotted to each eye. Higher score will indicate severity of the disease (dry eye).
  Tear osmolarity OU was assessed using the TearLab Osmolarity System Test by collecting nanoliter volumes of tear fluid at each visit from each eyelid margin using the Osmolarity Test Pen and Test Card. Results were interpreted according to the provided instructions and scores (mOsm/L) for each eye were recorded. Normal, mild/moderate, and severe dry eyes had average tear osmolarity values of approximately 302+/-8 mOsm/L, 315+/-10 mOsm/L and 336+/022 mOsm/L, respectively.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mOsm/L
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 125
mOsm/L
  OD- Right eye | -4.0 (19.44)
  OS- left eye | -11.7 (18.54)
Statistical Analysis 1: Comparison: CequaTM (Cyclosporine 0.09%) Ophthalmic Solution; Test type: Other — Single group analysis; p = 0.0323, Paired t-test; OD- Right eye p value
Statistical Analysis 2: Comparison: CequaTM (Cyclosporine 0.09%) Ophthalmic Solution; Test type: Other — Single group analysis; p = 0.3447, Paired t-test — OS: P-Value

6. Secondary Outcome: Mean Change From Baseline in Frequency of Artificial Tear Product Use.
Description: Based on entries in the subject diaries, frequency of artificial tear product use will be assessed.
  Frequency for artificial tear: This is number of times per day recorded in a daily diary log assessed at baseline and week 12. The higher the number the worse the outcome. The lower the number the better the outcome
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: times product used/day
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 124
times product used/day | -1.5 (2.39)
Statistical Analysis 1: Comparison: CequaTM (Cyclosporine 0.09%) Ophthalmic Solution; Test type: Other — Single group analysis; p < 0.0001, Paired t-test

7. Secondary Outcome: Schirmer's Test Score
Description: An unanesthetized Schirmer's test was performed in each eye at least 5 minutes after the lissamine green conjunctival staining to allow for any reflex tearing to subside. At each visit, strips were placed OU at the same time and timed for 5 min. Strips were removed after 5 min and the amount of wetting was recorded in mm and also marked with a line on the strip. The Investigator recorded a score for each eye. A score of greater than 10 mm in 5 minutes is accepted as normal. A score of less than 5 mm in 5 minutes indicates a tear deficiency. A score less than 10 mm in 5 minutes indicates a change from normal in tear production.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 125
mm | 2.4 (8.61)
Statistical Analysis 1: Comparison: CequaTM (Cyclosporine 0.09%) Ophthalmic Solution; Test type: Other — Single group analysis; p = 0.0029, Paired t-test

8. Secondary Outcome: Percentage of Subjects Who Prefer Study Treatments Over Prior Treatment.
Description: Subjects will be asked, which treatment they prefer for the management of the dry eye (prior treatment or study treatment).
  Note- For this outcome measure, participants were provided the option to not choose either treatment as the preferred treatment.
Time Frame: Week 12
Measure: Number; unit: percentage of participants
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
Number analyzed (Participants) | 113
percentage of participants
  Prefer prior treatment | 21.8
  Prefer study treatment | 69.4

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/134
Serious Adverse Events (participants affected / at risk) | 0/134
Other Adverse Events (participants affected / at risk) | 20/134
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CequaTM (Cyclosporine 0.09%) Ophthalmic Solution (N=134)
Instillation Site Irritation (General disorders) | 17
Instillation Site Pain (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT04357795/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT04357795/SAP_001.pdf